CLINICAL TRIAL: NCT01601873
Title: A Randomized Controlled Comparative Study on Efficacy and Cost-effectiveness of Heparin-bonded Versus Non-heparin-bonded Polytetrafluroethylene Hemodialysis Access Grafts.
Brief Title: Propaten Randomized Investigation on Cost-benefit and Efficacy
Acronym: PRICE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Results from futility analysis conducted at planned interim time-point did not meet the study criteria for continuation.
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: University Hospitals Cleveland Medical Center (Other); University of Arkansas (Other); Ochsner Health System (Other)
Responsible Party: Principal Investigator, Kristofer Charlton-Ouw, Associate Professor, Department of Cardiothoracic and Vascular Surgery, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTVS-KC01; UTHSCMS-12/0095 (Other: UTHSC IRB)
Record Dates: First submitted 2012-05-16; First posted 2012-05-18 (Estimated); Results first posted 2019-02-27 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-01

CONDITIONS: End-stage Renal Disease
Keywords: Arteriovenous graft; Propaten; Heparin-bonded; hemodialysis vascular access; Surgical; Arteriovenous Shunt
MeSH Terms: conditions — Kidney Failure, Chronic; Arteriovenous Fistula

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- PROPATEN (Experimental): patients with heparin-bonded graft implantation
  Interventions: Device: PROPATEN
- Standard Graft (Active Comparator): patients undergoing ePTFE hemodialysis graft implantation
  Interventions: Device: Standard Graft

INTERVENTIONS:
Device: PROPATEN — Heparin-bonded graft implantation for hemodialysis vascular access
  Other Names: Heparin-bonded hemodialysis graft
  Arms: PROPATEN
Device: Standard Graft — non-heparin bonded conventional hemodialysis vascular access graft
  Other Names: Conventional ePTFE hemodialysis graft
  Arms: Standard Graft

SUMMARY:
The purpose for this study is to evaluate the patency and outcomes of conventional and heparin anticoagulant bonded arteriovenous grafts in patients with end stage renal disease.

DETAILED DESCRIPTION:
Study Design: This is a prospective, multi-institution, parallel-group, single-blinded, randomized-controlled, two-arm, effectiveness study comparing heparin-bonded (Propaten®) versus non-heparin-bonded arteriovenous grafts.

Procedure: In patients without usable native vein, prosthetic arteriovenous grafts will be implanted for hemodialysis access. Patients will be randomized intraoperatively to either conventional (Gore® Stretch) or heparin-bonded grafts (Gore® Propaten).

Course of Study: The study will accrue patients over the course of 5 years.

Enrollment: Enrollment will consist of adult patients who require hemodialysis. If the patient cannot have a native vein arteriovenous fistula, the patient is a candidate for arteriovenous graft. Patients will be screened and consented preoperatively. If the intraoperative decision is made that the patient will require a graft, randomization will occur and the patient will be considered enrolled.

Recruitment: The target population comprises of all adult patients aged 18 years and above with end stage renal disease requiring arteriovenous access for hemodialysis. The target for enrollment will be 200 patients.

Risks: The standard or known adverse events associated with graft implantation include thrombosis, infection, pseudoaneurysm, hematoma, and venous stenosis. There are case reports of heparin sensitivity. The investigators do not expect any additional physical risks other than an unintentional disclosure of sensitive patient health information.

Data Safety Monitoring: As the Principal Investigator of this study, Dr. Charlton-Ouw from the Department of Cardiothoracic and Vascular Surgery at The University of Texas at Houston Medical School will conduct the data safety monitoring of this study. He will annually meet with all other co-investigators to review the patients enrolled in this study. As part of the data safety monitoring plan, all patients enrolled until that point in time would be unblinded in order to review the outcomes. Interim analyses will be conducted at the one-year follow up time.

IND#: The devices that will be used are already approved by the FDA and do not have IND#.

Proposed Funding Source: The study is internally funded.

Communication of Study Results: The communication of study results will occur only between authorized individuals who are listed to take part in the study through our department. The individuals who will take part in the study will acknowledge and adhere to the importance of patient safety and the protection of their private information. The results of this study will be analyzed and published after the approval of the principal investigator, co-investigators, and biostatistician in a peer-reviewed scientific journal and/or presented at an international/national scientific conference or meeting regardless of outcome.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years of all ethnicities
* End-stage Renal Disease stage 4 (GFR 15-29 ml/min 1.73m2) or stage 5 (GFR <15ml/min 1.73m2) per National Kidney Foundation guidelines
* Currently undergoing hemodialysis with a failure of previous access
* Expected to undergo hemodialysis within 6 months of presentation

Exclusion Criteria:

* Unable/refuse to abide with follow-up
* Known hypercoagulability syndrome or a bleeding disorder
* On a previous anticoagulant treatment
* Intraoperative decision in favor of fistula instead of graft
* Pregnant or breast-feeding women
* A documented history of heparin induced thrombocytopenia or allergy
* Active infections
* Evidence or suspicion of central vein stenosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2012-11-09 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristofer M Charlton-Ouw, MD, Principal Investigator — University of Texas Health Science Center, UT Medical School Department of Cardiothoracic and Vascular Surgery, Houston
Locations (5):
- United States (5):
  - University of Arkansas for Medical Sciences (UAMS) & Central Arkansas Veterans Healthcare System (CAVHS), Little Rock, Arkansas
  - John Ochsner Heart & Vascular Institute Ochsner Medical Center, New Orleans, Louisiana
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Department of Cardiothoracic and Vascular Surgery and Memorial Hermann Heart and Vascular Institute - Texas Medical Center, Houston, Texas
  - Department of Cardiothoracic and Vascular Surgery; Memorial Hermann Hospital Southeast, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided
De-identified data will be available following institutional review board approval

REFERENCES:
- [Background] Charlton-Ouw KM, Nosrati N, Miller CC 3rd, Coogan SM, Safi HJ, Azizzadeh A. Outcomes of arteriovenous fistulae compared with heparin-bonded and conventional grafts for hemodialysis access. J Vasc Access. 2012 Apr-Jun;13(2):163-7. doi: 10.5301/JVA.2011.8715. PMID 21983827

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 103 were enrolled, but only 97 started (a difference of 6 subjects). These 6 subjects who were enrolled but did not start the study presented to the day-surgery operating room but had not followed instructions to stop Coumadin; therefore, their cases were cancelled.
Period: Overall Study
Arm/Group | PROPATEN | Standard Graft
Started | 50 | 47
Completed | 48 | 44
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PROPATEN | Standard Graft | Total
Number analyzed (Participants) | 50 | 47 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (12.6) | 65 (11.9) | 64.6 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 21 | 51
  Male | 20 | 26 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 5 | 14
  Not Hispanic or Latino | 41 | 42 | 83
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50 | 47 | 97

OUTCOME MEASURES:

1. Primary Outcome: Primary Graft Patency Rate
Description: Primary graft patency refers to the successful use of a vascular access for hemodialysis without any surgical or endovascular intervention.
Time Frame: 12 months
Population: 1 in the propaten arm and 3 in the standard graft arm were lost to follow up.
Measure: Number; unit: Percentage of participants
Arm/Group | PROPATEN | Standard Graft
Number analyzed (Participants) | 49 | 44
Percentage of participants | 35 | 33
Statistical Analysis 1: Comparison: PROPATEN vs Standard Graft; Test type: Superiority; p = 0.884, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Primary-Assisted Graft Patency Rate
Description: Primary-assisted graft patency is defined as a patent access with evidence of malfunction that requires an open surgical or endovascular intervention.
Time Frame: 12 months
Population: 1 in the propaten arm and 3 in the standard graft arm were lost to follow up.
Measure: Number; unit: Percentage of participants
Arm/Group | PROPATEN | Standard Graft
Number analyzed (Participants) | 49 | 44
Percentage of participants | 57 | 60
Statistical Analysis 1: Comparison: PROPATEN vs Standard Graft; Test type: Superiority; p = 0.946, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Secondary Graft Patency Rate
Description: Secondary graft patency is defined as a functional access following intervention for thrombosis or after any interposition grafting for any reason including stenosis, aneurysm or pseudoaneurysm.
Time Frame: 12 months
Population: 1 in the propaten arm and 3 in the standard graft arm were lost to follow up.
Measure: Number; unit: Percentage of participants
Arm/Group | PROPATEN | Standard Graft
Number analyzed (Participants) | 49 | 44
Percentage of participants | 62 | 52
Statistical Analysis 1: Comparison: PROPATEN vs Standard Graft; Test type: Superiority; p = 0.294, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Primary Graft Patency Rate
Description: as for outcome 1
Time Frame: 24 months after graft placement
Population: 2 in the propaten group and 3 in the standard graft group were lost to follow up.
Measure: Number; unit: Percentage of participants
Arm/Group | PROPATEN | Standard Graft
Number analyzed (Participants) | 48 | 44
Percentage of participants | 24 | 25
Statistical Analysis 1: Comparison: PROPATEN vs Standard Graft; Test type: Superiority; p = 0.538, Log Rank

5. Primary Outcome: Primary-Assisted Graft Patency Rate
Description: as for outcome 2
Time Frame: 24 months after graft placement
Population: 2 in the propaten group and 3 in the standard graft group were lost to follow up.
Measure: Number; unit: Percentage of participants
Arm/Group | PROPATEN | Standard Graft
Number analyzed (Participants) | 48 | 44
Percentage of participants | 26 | 22
Statistical Analysis 1: Comparison: PROPATEN vs Standard Graft; Test type: Superiority; p = 0.786, Log Rank

6. Primary Outcome: Secondary Graft Patency Rate
Description: as for outcome 3
Time Frame: 24 months after graft placement
Population: 2 in the propaten group and 3 in the standard graft group were lost to follow up.
Measure: Number; unit: Percentage of participants
Arm/Group | PROPATEN | Standard Graft
Number analyzed (Participants) | 48 | 44
Percentage of participants | 48 | 38
Statistical Analysis 1: Comparison: PROPATEN vs Standard Graft; Test type: Superiority; p = 0.185, Log Rank

7. Secondary Outcome: Number of Participants With Complications or Morbidity Attributable to the Study
Description: Complication/morbidity associated with both types of interventions
Time Frame: at least 1 year but up to two years
Population: 2 in the propaten group and 3 in the standard graft group were lost to follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | PROPATEN | Standard Graft
Number analyzed (Participants) | 48 | 44
Participants | 0 | 0

8. Secondary Outcome: Cost Estimation and Analysis
Description: Will be based on the difference between total cost analysed on the basis of the specific graft price, cost of re-intervention procedures if any, treatment of complications, hospital stay, etc., and compared for each study arm.
Time Frame: During the study period based on an average participant follow-up of 2 years after graft placement
Population: The cost data were not collected.
Arm/Group | PROPATEN | Standard Graft
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Quality of Life (QoL) Comparison
Description: Comparative assessment of quality of life reported by the patients in two arms
Time Frame: Participants would be followed for a period of 2 years after graft placement
Population: Qol data was collected, but because results of a planned interim futility analysis did not meet the study criteria for continuation, we do not believe analysis of the QoL data would be meaningful. Analysis of QoL data is an extremely onerous process that would take months to conduct. It is not worth the resources required to perform this analysis.
Arm/Group | PROPATEN | Standard Graft
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Number of Postoperative Re-interventions
Time Frame: at least 1 year but up to two years
Population: 2 in the propaten group and 3 in the standard graft group were lost to follow up.
Measure: Mean (Standard Deviation); unit: post-operative re-interventions
Arm/Group | PROPATEN | Standard Graft
Number analyzed (Participants) | 48 | 44
post-operative re-interventions | 2.7 (5.0) | 2.0 (2.5)

ADVERSE EVENTS:
Time Frame: At least 1 year but up to two years (the study was stopped early for futility; therefore, some subjects were only followed for a year)
Arm/Group | PROPATEN | Standard Graft
All-Cause Mortality (participants affected / at risk) | 7/48 | 4/44
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/44
Other Adverse Events (participants affected / at risk) | 19/48 | 20/44
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PROPATEN (N=48) | Standard Graft (N=44)
stenosis (Vascular disorders) | 7 (7) | 8 (8)
Unable to cannulate (Surgical and medical procedures) | 7 (7) | 5 (5)
Graft site bleeding (Surgical and medical procedures) | 2 (2) | 0 (0)
Vascular steal requiring intervention (Vascular disorders) | 3 (3) | 3 (3)
Pseudoaneurysm (Vascular disorders) | 0 (0) | 2 (2)
Failure to mature (Vascular disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
The trial was stopped early for futility based on a pre-planned interim analysis and a Bayesian probability forecast incorporating all available information from a recent meta-analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-14): https://cdn.clinicaltrials.gov/large-docs/73/NCT01601873/Prot_SAP_000.pdf